CLINICAL TRIAL: NCT02402751
Title: Development, Implementation and Initiation of Normative Database Quantitative Ultra High Field MRI Paramaters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A0012148
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acquisition of normative database (Experimental): Development, implementation and initiation of normative database (image and data) quantitative ultra high field MRI paramaters
  Interventions: Procedure: acquisition of normative database with ultra high field MRI; Device: MRI

INTERVENTIONS:
Procedure: acquisition of normative database with ultra high field MRI — characterize non-invasively with an unprecedented resolution and sensitivity (high field MRI), anatomy as well as certain physiological, hemodynamic and metabolic function of brain, spinal cord, musculoskeletal system, and heart
Device: MRI

SUMMARY:
The Centre for Magnetic Resonance in Biology and Medicine (CRMBM, UMR-CNRS 7339 AMU) obtained funding for a whole body NMR imaging at 7. It is the only MRI at 7T installed in a hospital in France (only two 7T MRI in France) and therefore a unique opportunity to develop new diagnostic approaches.

The purpose of this study is to develop, implement and validate new MRI quantitative parameters derived from ultra high field MRI in order to characterize non-invasively with an unprecedented resolution and sensitivity, anatomy as well as certain physiological, hemodynamic and metabolic function of brain, spinal cord, musculoskeletal system, and heart in healthy subjects

DETAILED DESCRIPTION:
The key is that the goal of our projects is not only producing images of better quality than using a 3T scanner but also making images differently, by highlighting new contrasts and features of theses organs in order to improve the diagnosis and prognosis of neurological, psychiatric, cardiovascular and rheumatologic diseases.

ELIGIBILITY:
Inclusion Criteria:

* People not presenting contraindications to the MRI (pacemaker, agitation, metallic brightness, claustrophobia etc.)
* People having no intra-physical object potentially conductive.
* People having no affection after detailed interrogation

Exclusion Criteria:

* People staying in a sanitary or social establishment
* People in emergency situation
* People not wishing to be informed about anomalies in the MRI
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
qualitative validation concerning structure visible with high field MRI | 4 years
  the validation criteria are qualitative (contrast and visibility of anatomical structures usually visible 7T but not visible at 3T will be used to assess the sensitivity of images for each modality) and quantitative (signal to noise ratio (SNR), spatial and temporal resolution).

SECONDARY OUTCOMES:
acquisition of normative data and verification of the quality criteria obtained during the first phase | 4 years
  During the second phase, we will acquire normative data and verify the quality criteria of the first phase. Each quantitative variable will be extracted. After the acquisition of the first 30 volunteers for each parameter, the variance will be analyzed to assess the population distribution. Depending on the results, and issues raised by clinical research studies, other populations will be acquired

CONTACTS AND LOCATIONS:
Overall Officials: Maxime GUYE, M.D, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France